CLINICAL TRIAL: NCT00003236
Title: Randomized Phase II Study of Human C-raf Kinase Antisense Oligonucleotide Isis 5132 (CGP 69846A) or Human Pkc-Alpha Antisence Oligonucleotide ISIS 3521 (CGP 64128A) in Women With Previously Treated Matastatic Breast Cancer
Brief Title: Chemotherapy in Treating Women With Previously Treated Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066108; ECOG-3197
Record Dates: First submitted 1999-11-01; First posted 2004-06-09 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ISIS 3521; ISIS 5132

INTERVENTIONS:
Biological: ISIS 3521
Drug: ISIS 5132

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Randomized phase II trial to compare the effectiveness of ISIS 5132 with ISIS 3521 in treating women who have metastatic breast cancer that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the proportion of women with previously treated metastatic breast cancer who are progression free at 4 months after receiving ISIS 5132 or ISIS 3521. II. Determine duration of response to these treatment regimens in this patient population. III. Evaluate toxicities and tolerability of these treatment regimens in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to number of prior therapies for metastatic breast cancer (1 vs 2). Patients are randomized to one of two treatment arms. (Arm I closed 12/22/99) Arm I: Patients receive ISIS 5132 IV continuously over 21 days. (closed 12/22/99) Arm II: Patients receive ISIS 3521 IV continuously over 21 days. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity. After every 2 courses, patients are evaluated for response. Patients are followed every 3 months for the first 2 years, every 6 months the next 3 years, then annually thereafter.

PROJECTED ACCRUAL: A maximum of 68 patients (34 per arm) will be accrued in this study (Arm I closed 12/22/99).

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic adenocarcinoma of the breast Must have failed at least one but no more than two prior therapies for metastatic breast cancer, including endocrine and chemotherapy Relapsing while receiving or within 6 months of completing adjuvant chemotherapy Disease progression during or subsequent to the most recent therapy Measurable and evaluable disease Bone is an evaluable site only No CNS metastases Hormone receptor status: Estrogen receptor negative, positive, or unknown

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: Any status Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL AST/ALT less than 3 times upper limit of normal PTT within normal limits Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No active congestive heart failure No poorly controlled hypertension At least 3 months since prior myocardial infarction Other: No history of other malignant neoplasms, except curatively treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix Not pregnant or nursing Negative pregnancy test, documented sterilization, or postmenopausal status Fertile patients must use effective contraception No uncontrolled nonmalignant systemic diseases (including active peptic ulcer and poorly controlled diabetes mellitus) No underlying disease state associated with active bleeding No unexplained abnormality of prothrombin time (e.g., warfarin therapy)

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 28 days since prior chemotherapy Endocrine therapy: See Disease Characteristics At least 28 days since prior hormonal therapy Radiotherapy: Not specified Surgery: At least 2 weeks since major surgery Other: At least 28 days since prior use of other investigational drugs No therapeutic anticoagulation with heparin

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-07-13 (Actual); Primary Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J. Gradishar, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (6):
- United States (6):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Gradishar WJ, O'Neill A, Cobleigh M, et al.: A phase II trial with antisense oligonucleotide ISIS 3521/Cgp 64128a in patients (Pts) with metastatic breast cancer (MBC): ECOG trial 3197. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-171, 2001.